CLINICAL TRIAL: NCT07308496
Title: Computed Tomography-derived Fractional Flow Reserve vs. Angiographic Quantitative Flow Ratio in Management of Patients With Coronary Artery Disease
Acronym: CONQUER
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Collaborators: Fuwai Yunnan Cardiovascular Hospital (Other); Central China Fuwai Hospital of Zhengzhou University (Other); Shenzhen Sun Yat-sen Cardiovascular Hospital (Other); Ruijin Hospital (Other); Nanjing First Hospital, Nanjing Medical University (Other); The First Affiliated Hospital with Nanjing Medical University (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); The First Affiliated Hospital of Dalian Medical University (Other); Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025-2855
Record Dates: First submitted 2025-12-13; First posted 2025-12-29 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-12

CONDITIONS: Coronary Artery Disease
Keywords: CT-derived fractional flow reserve; Angiography-derived quantitative flow ratio
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- CT-FFR group (Experimental): The decisions of invasive angiography and revascularization will be guided by CT-FFR.
  Interventions: Diagnostic Test: CT-FFR guided strategy
- QFR group (Active Comparator): The decision of invasive angiography will be made as usual care, and revascularization will be guided by QFR.
  Interventions: Diagnostic Test: QFR guided strategy

INTERVENTIONS:
Diagnostic Test: CT-FFR guided strategy — Patients in this group will undergo CT-derived fractional flow reserve (CT-FFR) analysis. If the CT-FFR value is ≤0.80, patients will subsequently undergo invasive coronary angiography (ICA) and receive coronary revascularization. If the CT-FFR values of all vessels are >0.80, patients will not undergo invasive angiography.
  Arms: CT-FFR group
Diagnostic Test: QFR guided strategy — Patients in this group will undergo invasive coronary angiography (ICA) according to routine clinical indications. During the procedure, quantitative flow ratio (QFR) analysis will be performed. If the QFR value is ≤0.80, coronary revascularization will be performed. If the QFR value is >0.80, coronary revascularization will be forwent.
  Arms: QFR group

SUMMARY:
This is a multi-center, randomized controlled trial to compare the clinical outcomes between CT-derived fractional flow reserve (CT-FFR) guided strategy and angiography-derived quantitative flow ratio (QFR) guided strategy among patients with coronary artery disease (CAD). Participants who have at least one coronary stenosis of 70%-90% (vessel diameter ≥2.5 mm) detected by coronary CT angiography will be enrolled and are randomly assigned in a 1:1 ratio to CT-FFR guided group or QFR guided group. In CT-FFR group, the decisions of invasive angiography and revascularization will be guided by CT-FFR. In QFR group, the decision of invasive angiography will be made as usual care, and revascularization will be guided by QFR. The primary endpoint is the 1-year incidence of major adverse cardiac events (MACEs), including death, myocardial infarction, and unplanned revascularization.

ELIGIBILITY:
Patient-level inclusion criteria:

1. Adults aged ≥18 years.
2. Patients with stable angina, unstable angina, or post-myocardial infarction ≥72 hours.
3. Patients are able and willing to provide written informed consent.

Lesion-level inclusion criteria:

(1) Coronary CT angiography (CCTA) shows at least one coronary artery with 70%-90% diameter stenosis and vessel diameter ≥2.5 mm.

Patient-level exclusion criteria:

1. Previous percutaneous coronary intervention (PCI) or coronary artery bypass grafting (CABG).
2. Suspected acute myocardial infarction (ECG or biomarkers indicating acute phase).
3. Moderate to severe chronic kidney disease, defined as serum creatinine >150 μmol/L or estimated glomerular filtration rate (eGFR) <45 mL/min/1.73 m².
4. Severe valvular heart disease, aortic disease, or large ventricular aneurysm requiring surgery.
5. Atrial fibrillation or other severe cardiac arrhythmias.
6. Refusal or inability to sign informed consent.

Lesion-level exclusion criteria:

1. Poor-quality CCTA images that prevent CT-FFR analysis.
2. Severe coronary vessel tortuosity, overlapping segments, or other factors expected to cause poor-quality invasive angiography, hindering QFR measurement.
3. Combined with chronic total occlusion lesions.
4. The stenosis degree of the left main coronary artery was ≥50%.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1402 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Major Adverse Cardiac Events (MACEs) within 12 Months Post-Procedure | 12 Months Post-Procedural Follow-Up
  MACEs is defined as a composite of all-cause death, myocardial infarction, and unplanned revascularization.

SECONDARY OUTCOMES:
All-cause death | 12 Months After Randomization
  Death from any cause during the follow-up period.
Cardiac death | 12 Months After Randomization
  Death due to myocardial infarction, heart failure, or other cardiac causes.
Myocardial infarction (MI) | 12 Months After Randomization
  Defined according to the Fourth Universal Definition of Myocardial Infarction.
Repeat revascularization | 12 Months After Randomization
  Any planned or unplanned revascularization of the target vessel or graft.
Rehospitalization | 12 Months After Randomization
  Any hospital readmission for cardiac causes, recurrent angina, or other medical reasons.
Rate of invasive coronary angiography avoidance | 12 Months After Randomization
  The proportion of patients who avoided invasive coronary angiography after CT-FFR-based evaluation without adverse clinical outcomes.
Revascularization rate | 12 Months After Randomization
  The proportion of patients undergoing any coronary revascularization (PCI or CABG).
Number of stents implanted or bypass grafts performed | 12 Months After Randomization
  to assess procedural extent and resource utilization
Rate of optimal medical therapy | 12 Months After Randomization
  The proportion of patients treated conservatively without revascularization.
PCI rate | 12 Months After Randomization
  The proportion of patients receiving percutaneous coronary intervention.
CABG rate | 12 Months After Randomization
  The proportion of patients undergoing coronary artery bypass grafting.
Total cost | 12 Months After Randomization
  Including outpatient and inpatient diagnostic and treatment expenses, index hospitalization cost.

IPD SHARING:
Plan to Share IPD: No